CLINICAL TRIAL: NCT04446676
Title: Impact of the Type of Stabilization in the Two-stage Knee Reimplantation on Reinfection - Prospective, Randomized Study.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof A Gruca Teaching Hospital (Other)
Responsible Party: Principal Investigator, Bartosz Paweł, M.D., Ph.D., Prof A Gruca Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gruca Teaching Hospital
Record Dates: First submitted 2020-06-21; First posted 2020-06-25 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Knee Infection
Keywords: knee arthroplasty; infection; two-stage; sleeve; stem
MeSH Terms: conditions — Infections | interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Intervention Model Description: Two groups with endoprosthesis stabilisation with stem or sleeve.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stem stabilization (Active Comparator): Group of patients with stem endoprosthesis stabilization
  Interventions: Device: stabilization with stem
- Sleeve stabilization (Active Comparator): Group of patients with sleeve endoprosthesis stabilization
  Interventions: Device: stabilization with sleeve

INTERVENTIONS:
Device: stabilization with stem — In both groups revision endoprosthesis of knee will be implanted with stem or sleeve stabilization.
  Arms: Stem stabilization
Device: stabilization with sleeve — In both groups revision endoprosthesis of knee will be implanted with stem or sleeve stabilization.
  Arms: Sleeve stabilization

SUMMARY:
Participants after first-stage of knee infection reimplantation will be assign to one of two groups: with stem vs. with sleeve. Investigators will check participants on clinical, laboratory and reinfection signs. The main hypothesis is that better mechanical stability of endoprosthesis with sleeves will support infection treatment.

DETAILED DESCRIPTION:
All participants will be treated because of periprosthetic joint infection of the knee, after primary arthroplasty. All participants will be treated with two-stage protocol. In first stage debridement and spacer implantation will be performed. After 6-week antibiotics, when will be absent clinical or laboratory signs of reinfection, second stage will be performed. All participants upon fulfillment all inclusion and exclusion criteria will sign informed consent. With computer software patients will be randomized to one of two groups: with stem vs. with sleeve. After operation all patients will get target antibiotics for 3 weeks. Pre-operation and after on periodic controls will checked the Knee Society Score, The Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC), Visual Analogue Scale. After 2-year observation evaluation of reinfection rate will be performed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* second-stage of knee reimplantation
* primary knee replacement in primary knee osteoarthritis
* fulfillment of International Consensus Meeting 2018 infection criteria

Exclusion Criteria:

* intraoperative bone defects Anderson Orthopedic Research Institute score >II
* autoimmune disease
* diabetes
* peripheral vascular disease
* congenital or acquired immunodeficiencies
* lack of pathogens after first-stage
* multi-bacterial infection
* multidirectional instability
* lack of patient consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Reinfection | 2 years
  Rate of reinfection in both groups

SECONDARY OUTCOMES:
Loosening radiological signs | 2 years
  Radiological evaluation of implant loosening with Modern Knee Society Radiographic Evaluation System

OTHER OUTCOMES:
Knee Society Score | 1 year
  Clinical evaluation of patients after knee revision
The Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) | 1 year
  Clinical evaluation of patients after knee revision
Visual Analogue Score | 1 year
  Clinical evaluation of patients after knee revision
Alignment | 6 weeks
  Radiological alignment of knee after operation in degrees
C-reactive protein | 1 year
  After operation and at period controls (mg/l)
Erythrocyte sedimentation rate | 1 year
  After operation and at period controls (mm/h)

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Bartosz, Principal Investigator — Prof. A. Gruca Teaching Hospital in Otwock
Locations (1):
- Gruca Teaching Hospital, Centre of Postgraduate Medical Centre, Otwock, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and Informed consent form will be shared
Supporting Information: Study Protocol, ICF
Time Frame: 1 year